CLINICAL TRIAL: NCT04142671
Title: Determining Individualised Gait Modification Strategies to Reduce Knee Joint Moments in Alkaptonuria Patients Using Real-time Feedback
Brief Title: Individualised Gait Modification Strategies in Alkaptonuria Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Liverpool John Moores University (Other)
Collaborators: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Hannah Shepherd, Associate Lecturer in Clinical Biomechanics, Liverpool John Moores University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19LJMUSPONSOR086; 248641 (Other: IRAS Project ID)
Record Dates: First submitted 2019-10-24; First posted 2019-10-29 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Alkaptonuria
MeSH Terms: conditions — Alkaptonuria

STUDY DESIGN:
Intervention Model Description: Single group trial pre- post-intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individualised Gait Modification Intervention (Experimental): Patients will carry out several walking trials to test the efficacy of an individualised gait modification intervention.
  Pre-intervention over ground walking, pre-intervention treadmill walking, intervention treadmill walking with real-time biofeedback on their knee loading, intervention treadmill walking with no feedback, and post-intervention over ground walking.
  Interventions: Other: Individualised gait modification intervention

INTERVENTIONS:
Other: Individualised gait modification intervention — An individualised gait modification intervention to reduce knee joint loading. Knee joint loading will be presented in real-time during treadmill walking. A 10% reduction of each patients baseline knee loading will be used as a target threshold along with visualisation of the history of 5 previous steps. Patients are encouraged to determine their own gait modification strategy that is most efficient for them. Previous examples of gait modifications that mechanically reduce knee loading will be presented to them.

SUMMARY:
This study evaluates the efficacy of a gait modification intervention using real-time biofeedback on reducing the knee joint loading in Alkaptonuria patients during treadmill walking. It will also assess whether the individualised adopted gait modification can be retained without feedback and during over ground walking.

DETAILED DESCRIPTION:
Alkaptonuria (AKU) is a degenerative disease affecting the cartilage of the joints. The disease affects movement function, particularly walking/gait which is an important activity of daily living. It is believed that increased joint loading measured by the moments acting upon the joints, contributes to the degeneration of joint cartilage in Alkaptonuria, particularly in the weight bearing joints such as the knee and hips, resulting in accelerated progression of painful symptoms. Currently there is no cure for Alkaptonuria and the current management includes joint replacement surgery. Gait modification strategy interventions could be a non-invasive alternative which could delay the time to surgical interventions by reducing or altering joint loading and stalling the progression of disease.

The aims of this study are 1) to determine if individualised gait modification strategies can be used to reduce the 3D knee joint loading, 2) to determine if the gait modifications can be retained without feedback during over ground walking and 3) to determine the individualised gait modification strategies adopted by AKU patients.

Gait data will be measured and quantified using the non-invasive typical clinical gait analysis set up, using 3D motion capture combined with force data whereby joint angles, moments and powers can be calculated in all 3 planes of motion during treadmill walking. The intervention will involve real-time biofeedback using Motek's M-Gait treadmill. Due to the heterogeneity of the sample, each AKU patient will act as their own control. Gait data will be compared pre- and post-intervention and a validated pain score will be used to identify any patterns with knee pain and adopted gait modifications.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of Alkaptonuria
* Able to understand written and spoken English.
* Willing and able to give informed consent to participate
* Above the age of 18.

Exclusion Criteria:

* The reliance on or use of a walking aid.
* Any previous lower limb joint replacements.
* Any severe pain or unable to walk comfortably and consecutively for 20 minutes.
* Pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline 3D knee joint moment impulse after intervention | At baseline and immediately after the intervention
  This represents the knee joint load during walking measured from kinematic and kinetic data obtained during the 3D gait analysis

SECONDARY OUTCOMES:
Change from baseline joint angles after intervention | At baseline and immediately after the intervention
  Lower limb joint angles in degrees measured from kinematic data obtained during the 3D gait analysis
Change from baseline joint moments after intervention | At baseline and immediately after the intervention
  Lower limb joint moments in Nm/kg measured from kinematic and kinetic data obtained during the 3D gait analysis
Change from baseline joint powers after intervention | At baseline and immediately after the intervention
  Lower limb joint powers in Watts/kg measured from kinematic and kinetic data obtained during the 3D gait analysis
Knee injury and Osteoarthritis Outcome Score | Pre-intervention
  Validated Knee injury and Osteoarthritis Outcome Score Questionnaire. Scores between 0-100, 0 representing extreme problems and 100 representing no problems.

CONTACTS AND LOCATIONS:
Overall Officials: Gabor J Barton, MD, PhD, Study Director — Liverpool John Moores University

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers

REFERENCES:
- [Background] Simic M, Hinman RS, Wrigley TV, Bennell KL, Hunt MA. Gait modification strategies for altering medial knee joint load: a systematic review. Arthritis Care Res (Hoboken). 2011 Mar;63(3):405-26. doi: 10.1002/acr.20380. Epub 2010 Oct 27. PMID 20981808
- [Background] Taylor AM, Boyde A, Wilson PJ, Jarvis JC, Davidson JS, Hunt JA, Ranganath LR, Gallagher JA. The role of calcified cartilage and subchondral bone in the initiation and progression of ochronotic arthropathy in alkaptonuria. Arthritis Rheum. 2011 Dec;63(12):3887-96. doi: 10.1002/art.30606. PMID 22127706